CLINICAL TRIAL: NCT07044297
Title: A Phase 3, Randomized, Active-Controlled, Double-Blind Clinical Study to Evaluate the Efficacy and Safety of MK-8527 Oral Once-Monthly as HIV-1 Preexposure Prophylaxis
Brief Title: A Clinical Study of MK-8527 to Prevent Human Immunodeficiency Virus Type 1 (HIV-1) (MK-8527-011)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8527-011; MK-8527-011 (Other: MSD); 2025-520610-58-00 (Registry Identifier: EU CT); U1111-1317-6239 (Registry Identifier: UTN)
Record Dates: First submitted 2025-06-26; First posted 2025-06-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Human Immunodeficiency Virus (HIV); HIV Pre-Exposure Prophylaxis
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MK-8527 (Experimental): Participants will receive 11 mg MK-8527 once monthly (QM) and placebo to FTC/TDF once daily (QD) for up to approximately 2 years. Participants will then receive open-label 200 mg FTC/245 mg TDF QD for an additional 28 days.
  Interventions: Drug: MK-8527; Drug: FTC/TDF; Drug: Placebo to FTC/TDF
- FTC/TDF (Active Comparator): Participants will receive 200 mg FTC/245 mg TDF QD and placebo to MK-8527 QM for up to approximately 2 years. Participants will then receive open-label 200 mg FTC/245 mg TDF QD for an additional 28 days.
  Interventions: Drug: FTC/TDF; Drug: Placebo to MK-8527

INTERVENTIONS:
Drug: MK-8527 — Oral tablet
  Arms: MK-8527
Drug: FTC/TDF — Oral tablet
  Other Names: Truvada; Emtricitabine/Tenofovir Disoproxil Fumarate
Drug: Placebo to MK-8527 — Placebo tablet matched to MK-8527
  Arms: FTC/TDF
Drug: Placebo to FTC/TDF — Placebo tablet matched to FTC/TDF
  Arms: MK-8527

SUMMARY:
Researchers are looking for new medicines to prevent HIV-1 (Human Immunodeficiency Virus Type 1) infection.

The goals of this study are to learn:

* If taking MK-8527 once a month works to prevent HIV-1 infection as well as or better than a standard (usual) pre-exposure prophylaxis (PrEP) taken once a day
* About the safety of MK-8527 and if people tolerate it

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Is confirmed HIV-uninfected based on negative HIV-1/HIV-2 test results
* Is a cisgender man, transgender woman (assigned male sex at birth), transgender man (assigned female sex at birth), or gender nonbinary person
* Has had condomless receptive anal sex in the 12 months prior to screening (not including sex occurring in a mutually monogamous relationship) and has at least 1 of the following: receptive anal sex with 2 or more partners in the 3 months prior to screening (regardless of condom use), rectal or urethral gonorrhea or chlamydia or incident syphilis in the 6 months prior to screening, or any self-reported stimulant drug use with sex in the 3 months prior to screening
* Weighs ≥35 kg

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has hypersensitivity or other contraindication to any component of the study interventions
* Has evidence of acute or chronic hepatitis B infection
* Has a history of malignancy within 5 years of screening except for adequately treated basal cell or squamous cell skin cancer, or in situ anal or cervical cancers
* Has taken cabotegravir, lenacapavir, or any other long-acting HIV prevention product at any time
* Is receiving or is anticipated to require any prohibited therapies from 30 days prior to Day 1 through the study duration
* Has received an HIV vaccine at any time (ie, through past participation in an investigational clinical study) or monoclonal antibodies to HIV within 12 months before Day 1
* Is expecting to donate eggs at any time during the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4390 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2027-07-22 (Estimated); Study Completion 2027-07-22 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adjudicated Human Immunodeficiency Virus Type 1 (HIV-1) Infection | Up to approximately 2 years
  The number of participants with adjudicated HIV-1 infection will be determined.
Number of Participants Who Experience At Least One Adverse Event (AE) | Up to approximately 2 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants that experienced AEs will be reported.
Number of Participants Who Discontinue Study Intervention Due to an AE | Up to approximately 2 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants that discontinued study intervention due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (66):
- United States (23):
  - University of Alabama at Birmingham-UAB 1917 Research Clinic ( Site 0006), Birmingham, Alabama
  - USA Health University Hospitals ( Site 0020), Mobile, Alabama
  - UCLA Center for Clinical AIDS Research and Education ( Site 0004), Los Angeles, California
  - Bridge HIV - San Francisco Department of Public Health ( Site 0001), San Francisco, California
  - Whitman-Walker Institute ( Site 0016), Washington D.C., District of Columbia
  - University of Miami RAPID Research ( Site 0003), Miami, Florida
  - Orlando Immunology Center ( Site 0021), Orlando, Florida
  - Hope Clinic of the Emory Vaccine Center ( Site 0009), Decatur, Georgia
  - University of Illinois Chicago ( Site 0027), Chicago, Illinois
  - University Medical Center New Orleans ( Site 0024), New Orleans, Louisiana
  - Open Arms Healthcare Center ( Site 0025), Jackson, Mississippi
  - Rutgers New Jersey Medical School ( Site 0010), Newark, New Jersey
  - Montefiore Medical Center ( Site 0017), The Bronx, New York
  - NC TraCS Institute - CTRC; University of North Carolina at Chapel Hill ( Site 0008), Chapel Hill, North Carolina
  - Regional Center for Infectious Diseases ( Site 0018), Greensboro, North Carolina
  - Philadelphia Fight Community Health Centers ( Site 0011), Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center-Division of Infectious Diseases ( Site 0022), Pittsburgh, Pennsylvania
  - Prisma Health Richland Hospital-Clinical Research Unit ( Site 0007), Columbia, South Carolina
  - St. Jude Children's Research Hospital ( Site 0026), Memphis, Tennessee
  - Meharry Medical College ( Site 0013), Nashville, Tennessee
  - Central Texas Clinical Research ( Site 0014), Austin, Texas
  - Saint Hope Foundation, Inc. ( Site 0015), Bellaire, Texas
  - Fred Hutchinson Cancer Center - The Seattle HIV Vaccine Trials Unit ( Site 0002), Seattle, Washington
- Argentina (5):
  - Centro de Estudios Infectológicos S.A. ( Site 0357), CABA, Buenos Aires
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada ( Site 0352), CABA, Buenos Aires
  - Fundación Huésped ( Site 0350), CABA, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata ( Site 0353), Mar del Plata, Buenos Aires
  - Fundación IDEAA ( Site 0351), Buenos Aires
- Brazil (7):
  - Fundaçao de Medicina Tropical Doutor Heitor Vieira Dourado ( Site 0412), Manaus, Amazonas
  - Obras Sociais Irma Dulce ( Site 0406), Salvador, Estado de Bahia
  - School of Medicine Federal University of Minas Gerais ( Site 0417), Belo Horizonte, Minas Gerais
  - Hospital Geral de Nova Iguacu ( Site 0411), Nova Iguaçu, Rio de Janeiro
  - Ricardo Diaz Scientific Solutions ( Site 0402), São Paulo, São Paulo
  - Centro de Referência e Treinamento DST/AIDS ( Site 0400), São Paulo, São Paulo
  - Hospital das Clinicas FMUSP ( Site 0401), São Paulo, São Paulo
- Chile (3):
  - Universidad San Sebastian - Providencia ( Site 0454), Santiago, Region M. de Santiago
  - Universidad de Chile - Hospital Clínico Universidad de Chile-Inmunologia Alergia y VIH ( Site 0450), Santiago, Region M. de Santiago
  - Hospital Dr. Hernán Henríquez Aravena ( Site 0451), Temuco, Región de la Araucanía
- Colombia (4):
  - IPS SURA San Diego ( Site 0500), Medellín, Antioquia
  - Clinica de la Costa S.A.S. ( Site 0501), Barranquilla, Atlántico
  - Hospital Universitario San Ignacio ( Site 0503), Bogotá, Bogota D.C.
  - Fundación Valle del Lili ( Site 0502), Cali, Valle del Cauca Department
- Dominican Republic (3):
  - CEMDOE - Centro Médico de Diabetes, Obesidad y Especialidades ( Site 1001), Santo Domingo, Nacional
  - Endocardio ( Site 1003), Santo Domingo, Nacional
  - Instituto Dermatológico y Cirugía de Piel "Dr. Huberto Bogaert Díaz" ( Site 1002), Santo Domingo de Guzman, Santo Domingo Province
- France (3):
  - Hopital Saint Louis ( Site 0100), Paris
  - Hôpital Tenon ( Site 0102), Paris
  - Hopital Bichat - Claude Bernard ( Site 0101), Paris, Île-de-France Region
- Guatemala (3):
  - Clínica Médica Especializada en Pediatría e Infectología Pediátrica - Dr. Mario Melgar ( Site 1051), Guatemala City
  - MEDI-K ( Site 1053), Guatemala City
  - CELAN,S.A ( Site 1052), Guatemala City
- Universiti Malaya Medical Centre ( Site 0651), Kuala Lumpur, Malaysia
- Via Libre ( Site 0551), Lima, Peru
- South Africa (6):
  - Foundation For Professional Development ( Site 0257), King Williams Town, Eastern Cape
  - Wits RHI Research Center ( Site 0251), Johannesburg, Gauteng
  - Setshaba Research Centre ( Site 0252), Pretoria, Gauteng
  - Perinatal HIV Research Unit (PHRU) ( Site 0253), Soweto, Gauteng
  - Wits Maternal Adolescent and Child Health Research Unit (WMRU) ( Site 0256), Durban, KwaZulu-Natal
  - Desmond Tutu Health Foundation ( Site 0250), Cape Town, Western Cape
- Switzerland (3):
  - University Hospital Basel ( Site 1102), Basel, Canton of Basel-City
  - Inselspital Bern ( Site 1103), Bern, Canton of Bern
  - Checkpoint Zurich ( Site 1100), Zurich
- Thailand (4):
  - Chulalongkorn Hospital ( Site 0807), Bangkok, Bangkok
  - HIV Netherlands Australia Thailand Research Collaboration ( Site 0808), Bangkok, Bangkok
  - Faculty of Medicine Siriraj Hospital ( Site 0806), Bangkok, Bangkok
  - Research Institute for Health Sciences ( Site 0809), Muang, Chiang Mai

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com